CLINICAL TRIAL: NCT03864393
Title: Effect of a 12-week Multimodal Exercise Intervention on Walking Economy, Fatigability, and Propulsion in Individuals With Parkinson's Disease
Brief Title: Effect of Multimodal Exercise Training on Walking Economy in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POSSabilities
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
Keywords: walking economy; fatigability; propulsion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal overground locomotor training (Experimental): Individuals with Parkinson's Disease that meet the inclusion/exclusion criteria and enrolled in the study will participate in a 12-week multimodal exercise training intervention performed twice per week.
  Interventions: Other: Multimodal overground locomotor training

INTERVENTIONS:
Other: Multimodal overground locomotor training — Locomotor training sessions use various movement drills emphasizing power, stability, and stepping in a specific direction: forward, backward, lateral, rotational. Sessions also have an additional focus on gait initiation or steady-state walking. After circuit-style warm up exercises, participants perform overground movement drills that are specific to the emphasis of the individual training session, culminating in practicing everyday overground walking. Participants wear a heart rate monitor to ensure that the majority of the training session is performed at an aerobic intensity greater than 60% age predicted heart rate maximum (220-age +/- 5 bpm).

SUMMARY:
Sustained ambulation is a challenge for individuals with Parkinson's disease (PD) as walking economy is frequently compromised. There are also various disease-related skeletal muscle alterations that may contribute to performance fatigability during ambulation. Concomitantly, individuals with PD experience substantial difficulty maintaining sustained forward progression at push-off during the gait cycle due to diminished force production. Exercise is commonly prescribed for these individuals, though traditional exercise approaches to PD have often applied a "one impairment-one modality" paradigm that addresses each impairment separately. Interventions to optimize movement should facilitate an individual's response to the challenge of responding to a complex interplay of constraints that are also specific to a task and its environmental context. Thus, there are multiple concurrent targets for exercise interventions that may not fit easily within a "one impairment-one modality" model. A multimodal intervention is designed to address an array of constraining impairments concurrently. However, the evidence-base for multimodal exercise approaches is still developing and far from conclusive.

The purpose of this study is to demonstrate that multimodal overground locomotion training (OLT) can promote walking economy during sustained overground ambulation in individuals with PD, and produce concurrent secondary effects that decrease performance fatigability and increase propulsion. The aims of this study are to 1) Evaluate walking economy during sustained overground walking after 12 weeks of multimodal OLT, 2) Evaluate secondary effects of OLT.

DETAILED DESCRIPTION:
Protocol Overview: Subjects will be recruited from the greater Washington D.C. metro area. Individuals interested in participating as subjects will complete initial verbal screening to determine eligibility for inclusion. Those subjects who volunteer to participate will then be consented and enrolled for participation if exclusion and inclusion criteria are met.

Visit 1: (~120 minutes) Subjects will fill out a medical history form. Height and weight measurements will then be taken. The Hoehn and Yahr, Mini-Mental State Exam, Fatigue Severity Scale (FSS), Physical Activity Readiness Questionnaire (PAR-Q), and Physical Activity Scale in the Elderly (PASE) will then be administered. Subjects will first perform the 10-meter walk test. Subjects will be asked by researchers to walk 10 meters across a pressure sensitive walkway, 5 times at both comfortable speed and fast speed. After the 10-meter walk test, subjects will be given a 10-20 minute resting period before the second test. Subjects performing the 10-minute walk test will be fitted with a portable metabolic unit consisting of a face mask and torso apparatus. Wearable sensors will be secured to both arms, trunk, and legs. Before the test, subjects will stand in a resting position for at least 3 minutes to gain resting metabolic data. The subjects will then be asked to walk as far as they (the subjects) can in 10 minutes. Following the 10-minute walking period, subjects will again stand in a resting position to obtain recovery data. Subjects will then be given a 10-20 minute resting period during the transition to the third test. For the third test, subjects will be fitted with reflective markers at pre-specified anatomical landmarks used in a standardized gait marker set, for example medial and lateral knee and ankle joints. Electromyography (EMG) sensors will be placed on lower limb muscles. Subjects will then be asked to walk at both their preferred and fast walking speed over a 6 meter platform with embedded force plates. Subjects will be asked to perform as many trials as necessary to collect sufficient force plate data. After this test, subjects will be given the opportunity for a rest period if required before ending the testing day. For those subjects who start with the gait propulsion test, the testing order will include the same procedures yet in the reversed order.

Visit 2: (~90 minutes) Researchers will measure adipose tissue thickness over the calf muscle on the more affected leg (as indicated by the subject) using standard calipers. Subjects will then undergo a vascular occlusion test while resting in a semi-recumbent position. To perform this test investigators will place a large blood pressure cuff on the thigh and will place a NIRS optode on the calf muscle. Investigators will then inflate the cuff to 220mmHg to occlude blood flow to the lower leg. After a 5 minute period of occlusion the cuff pressure will be released and recovery NIRS data will be obtained. Subjects will then perform the CWRT Subjects will be fitted with 12-lead ECG and ICG sensors, will wear a face mask to collect metabolic data, and will be asked to perform the CWRT. Before the CWRT, subjects will rest for a minimum of 2 minutes in a standing position on a treadmill. During the CWRT subjects will be asked to walk at a constant speed for 6 minutes and 30 minutes with an 8 minute rest period between bouts. After the CWRT subjects will be asked to rest in a standing position to obtain recovery data. After this test, subjects will be given the opportunity to rest for a period if required before ending the testing day.

Visits 3-26: (~1 hour each) For these visits, subjects will perform an overground multimodal locomotor training protocol. Subjects will train individually with 1-2 trained instructors. Subjects will wear a Polar chest strap and a research grade pedometer during each session to enable instructors to modify training within the session to maintain a target intensity zone. The training protocol covers 12 weeks with two sessions per week for a total of 24 sessions.

Visit 27 (~90 minutes): Subjects will repeat the same testing procedures as they did in visit 1 in the same order as they did, determined by the initial randomization process.

Visit 28 (~90 minutes): Subjects will repeat the same testing procedures as they did in visit 2.

Study Procedures:

10-Meter Walk Test: The purpose of this test is to measure spatiotemporal variables related to walking at different speeds. Subjects will complete 10 repetitions of an over-ground 10-meter walk test on an instrumented pressure sensitive walkway. 5 repetitions will be performed at both comfortable and fast walking speeds.

10-Minute Walk Test (10MWT): The purpose of this test is to provide a method of perturbation for measuring both performance and perceived fatigability. Subjects will wear a fitted face mask and a torso unit as part of a portable metabolic unit. Wearable sensors will be secured on the torso, upper and lower limbs to measure gait characteristics. Subjects will rest in a standing position for at least 3 minutes prior to beginning this test to collect baseline data. Subjects will then walk as far as they can over a 10-minute interval or until they have to stop walking. Distance covered will be recorded at at 2.5-minute intervals throughout the test and at the end of the time walked if not the full 10 minutes. Velocity will be computed from the distances covered at the time intervals (meters/sec). The 10-minute walk test will be performed during the pre-intervention testing visit and post-intervention testing visit. Following the 10-minute walk period (or total time if ended early) subjects will rest in the standing position to obtain recovery data for at least 6 minutes.

Gait Propulsion Testing: Subjects will be outfitted with reflective markers comprised of a standardized full-body marker set for motion capture analysis. EMG sensors will be placed on muscle bellies of lower limb muscles. To establish the maximum voluntary contraction, subjects will be asked to contract muscles against resistance. Subjects will be asked to stand for system calibration for less than one minute and may be asked to move various limbs through a range of motion to ensure accuracy of the system prior to starting the test. Subjects will then be asked to walk across a 6-meter platform with embedded force plates enclosed by safety rails at their preferred and fast walking speed. Subjects will perform approximately 20-30 passes to ensure sufficient data collection by the force plates as appropriate contact with the force plate must be made for valid measurement. Once sufficient data has been collected, markers and sensors will be removed and the subject will be offered a seated rest period if needed.

Vascular Occlusion Test: During occlusion testing subjects will be seated in a semi-recumbent position on a plinth. A large blood pressure cuff will be fitted around the upper thigh with velcro straps to secure it in place. The cuff will be rapidly inflated in less than 5 seconds to above 220mmHg to restrict arterial and venous blood flow. The leg will be occluded for 5 minutes. The cuff pressure will then be released in less than 5 seconds and recovery variables will be recorded for an additional minimum of 3 minutes.

Constant Work Rate Treadmill Test (CWRT): During the CWRT subjects will be fitted with NIRS, Physioflow, and cardiopulmonary gas exchange devices to capture the cardiorespiratory measures. First, subjects will rest in a standing position for a minimum of 2 minutes. Second, treadmill will transition to the subjects' comfortable walking speed (average speed from the 10-meter walk test at comfortable speed). Third, after 6 minutes of continuous the treadmill will stop and subjects will rest for 8-minutes in a standing position. Fourth, after 8-minutes rest, the treadmill will transition to the subjects' comfortable walking speed and subjects will walk for a maximum of 30-minutes or until volitional exhaustion. Finally, subjects will recover for 10 minutes in a standing position. The speed used in the pre-test will be the same during the post-test

Multimodal Exercise Intervention: The intent of the multimodal training intervention is to encompass cardiovascular adaptations and locomotor improvements. To promote cardiovascular adaptation, training sessions will be adjusted in real-time to achieve a pre-determined target heart rate (HR) zone for each subject. HR will be monitored continuously during each training session. The target HR intensity during training sessions will be 60% of the subjects predicted maximal HR. The target HR zone will be 60% of predicated maximal HR +/- 5%. The subjects predicted maximal HR will be calculated using the formula: 220-age. Training procedures will include drills based on gait initiation and termination, agility, muscular power, and steady state actions. Drills will be conducted with an emphasis on direction change beyond usual forward progression. As subjects become familiar with the various drills, instructors will gradually increase the complexity, speed, and volume.

Propulsion Measures: For this study, propulsion will be defined by anterior peak positive ground reaction force (GRF) during overground walking. The force plates measure the GRF in response to the force placed upon it by the subject. In conjunction with motion capture analysis, the propulsive phase of gait can be determined and within that phase the anterior peak vector will be calculated. Peak propulsive force will be determined as the maxima (one point) of the anterior GRF.

Performance Fatigability Test Scoring: Performance fatigability is the rate or extent to which tissue, organ, system or total body function (fatigue) declines in response to a given task. After a 10-minute period of quiet rest in the sitting position, subjects will complete the 10-minute walk test. Distance covered will be recorded at the 2.5-minute interval of the test and for the total test. Velocities for the entire test (total distance walked / total minutes of test) and the first 2.5 minutes of the test (distance covered in the first 2.5 minutes / 2.5 minutes) will be calculated. The fractional change in velocity will then be computed as the quotient of total test velocity / 2.5 minute velocity. For example if the total test velocity and the 2.5-minute velocity were both 82 meters/minute, the total test velocity would be 100% of the velocity at 2.5 minutes. However, if the total test velocity were 80 meters/min and the velocity at 2.5 minutes were 82 meters/minute, then the total test velocity would be only .98 of the 2.5-minute velocity. To calculate the performance fatigability score, the fractional change in velocity will be divided by the distance covered. Thus any 2 subjects could have similar change in velocity scores (for example 0.5) but different total distances (100 versus 200 meters). In this case the performance fatigability score for the first subject would be 0.5/100 = 0.005 versus .5/200 = 0.0025. Scores are multiplied by 1000 to facilitate reporting. A small score indicates lower fatigability. Thus, even though the fractional change in velocity was similar for the 2 hypothetical subjects above, fatigability was less in the second subject as demonstrated by a lower performance fatigability score.

Perceived Fatigability Test Scoring: Perceived fatigability is the rate or magnitude of change in feelings of tiredness or weariness (symptoms of fatigue or perceived fatigue) in response to a given task. After the initial 10-minute sitting rest period, subjects will rate their perception of fatigue or vigor using the left side of the Fatigue and Fatigability Scale. Following the 10-minute walk test, subjects will be asked "compared to when you (the subject) started, how would you (the subject) rate your (the subject's) level of tiredness now" using the right side of the scale. The left side is considered a measure of fatigue because a change in fatigue was not assessed. The right side is considered to be a rating of fatigability because it assesses the change in tiredness. The score for the change in tiredness is then normalized to the total distance covered to calculate the perceived fatigability score: perceived fatigability = (change in tiredness / total distance walked) x 100 (multiplied by 100 to facilitate reporting and comparison).

Cardiopulmonary Gas Exchange Analyses: Gas exchange during the 10MWT will be collected using a wearable metabolic unit. The unit is calibrated prior to each test.

Cardiorespiratory Response to Treadmill Walking: Cardiorespiratory response during treadmill walking will be measured using NIRS, ICG, ECG, and pulmonary gas exchange devices. All measures are calibrated prior to each test.

Self-Reported Exertion During Treadmill Walking: During the CWRT subjects will be asked to rate their level of exertion using a Borg Scale.

Resting Skeletal Muscle Oxygenation and Hemodynamics: NIRS measurements of skeletal muscle oxygenation and hemodynamics will be recorded during the vascular occlusion test.

Motion capture system: Infrared cameras will capture movements of reflective markers worn by subjects within the volume. Reflective markers will be placed about the subject according to a predetermined full body gait marker model.

EMG sensors for measurement of muscle activity: EMG Electrodes are secured to the subject's skin over the muscle belly of interest. The sensor and electrode are covered with tape to minimize movement artifacts.

Force plates for GRF measurement: 4 force-plates are embedded in a 6 meter walkway. The force-plates measure x, y and z axes of the force and moment components, with the output signal fed into an amplifier.

Wearable sensors for measurement of gait characteristics: Wearable sensors contain accelerometers, gyroscopes, and magnetometers. Measurements are collected on the x, y, and z axes at a sample rate of 128 Hz. These sensors are attached to the preselected locations on the subject's body. This data is either wirelessly streamed via an access point and/or logged and stored in the sensor. Participants will also wear a step counter during each training sessions to record the total number of steps taken

Questionnaire:

Medical History Form: Subjects will fill out the medical history form on visit 1.

Testing/Forms:

Hoehn and Yahr: The Hoehn and Yahr scale (HY) is a widely used clinical rating scale, which defines broad categories of motor function in Parkinson's disease. This test will be administered by the researchers on visit 1.

Standardized Mini-mental State Exam: This test will be administered by researchers on visit 1 and is a 12-point questionnaire that addresses cognitive function.

Fatigue Severity Scale (FSS): This test will be administered by researchers on visit 1 and is a 9-item scale that measures the impact of fatigue on a person's activities and lifestyle.

Physical Activity Readiness Questionnaire (PAR-Q): This test will be administered by researchers on visit 1 and is a brief survey designed to screen individuals for potential contraindications for exercise participation.

Physical Activity Scale in the Elderly (PASE): This test will be administered by researchers on visit 1 and is a brief survey designed to assess physical activity in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosis of idiopathic Parkinson's Disease, mild to moderate (Hoehn and Yahr score less than or equal to 3)
* speaks English
* able to ambulate without requiring an assistive device

Exclusion Criteria:

* neurological disease diagnosis other than PD
* uncontrolled cardiovascular, pulmonary, neurological, or metabolic disease which may impact the ability to exercise or in which exercise is contraindicated
* any medications, such as beta-blockers, that may alter HR or metabolic data
* cognitive or psychiatric impairment precluding informed consent or ability to following instructions
* mini-Mental State Examination score <24
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Walking Economy | pre and post 12 week intervention protocol
  measured as oxygen consumption (VO2) over distance walked (meters) during a 10-minute walk test

SECONDARY OUTCOMES:
Change in Performance Fatigability | pre and post 12 week intervention protocol
  Performance fatigability severity is measured by the speed over the full time walked divided by speed in the first 2.5 minutes over total distance walked during the 10-minute walk test.
  Performance fatigability severity scores are multiplied by 1000 for reporting purposes. A higher score denotes greater fatigability.
  (Schnelle et al., 2012)
Change in Propulsion | pre and post 12 week intervention protocol
  Measured as peak anterior propulsive force measured using force plates during overground walking at the subject's preferred and fast walking speed.
Change in Interlimb Coordination | pre and post 12 week intervention protocol
  Interlimb coordination will be measured by phase relationship of limbs during overground walking
Change in Muscle Activation | pre and post 12 week intervention protocol
  EMG sensors will be placed on lower extremity muscles to measure the timing and amplitude of muscle activation throughout the gait cycle.
Change in Perceived Fatigability | pre and post 12 week intervention protocol
  Perceived fatigability severity is measured by dividing each subject's change in energy level pre and post 10-minute walk by the total distance walked (meters). Prior to starting the 10-minute walk subjects will be asked to rate their fatigue level using the left side of the scale (from 1-7: extremely energetic - extremely tired). After the 10-minute walk subjects will be asked to rate their change in energy level from the start of the test (1:extremely more energetic, 4:neither more tired nor energetic, 7:extremely more tired).
  Perceived fatigability severity scores are multiplied by 1000 for reporting purposes. A higher score denotes greater fatigability.
  (Schnelle et al., 2012)
Change in Cardiorespiratory Response to Treadmill Walking | pre and post 12 week intervention protocol
  Cardiorespiratory response to treadmill walking will be quantified by heart rate, VO2 consumption, VCO2 production, cardiac function, and peripheral muscle oxygen extraction during the CWRT.
Change in Self-Reported Exertion During Treadmill Walking | pre and post 12 week intervention protocol
  Self-reported exertion will be measured by asking subject to rate their level of perceived exertion using a Borg Scale during treadmill walking.
Change in Spatiotemporal Parameters during Overground Walking | pre and post 12 week intervention protocol
  Spatiotemporal parameters will be measured by stepping patterns during the over-ground 10-meter walk test.
Change in Resting Skeletal Muscle Oxygenation and Hemodynamics | pre and post 12 week intervention protocol
  Resting skeletal muscle oxygenation and hemodynamics of the calf muscle will be measured during the vascular occlusion test using a NIRS device.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Guccione, PT, PhD, DPT, Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnelle JF, Buchowski MS, Ikizler TA, Durkin DW, Beuscher L, Simmons SF. Evaluation of two fatigability severity measures in elderly adults. J Am Geriatr Soc. 2012 Aug;60(8):1527-33. doi: 10.1111/j.1532-5415.2012.04062.x. Epub 2012 Aug 2. PMID 22860899
- [Derived] Pugh RJ, Higgins RD, Min H, Wutzke CJ, Guccione AA. Turns while walking among individuals with Parkinson's disease following overground locomotor training: A pilot study. Clin Biomech (Bristol). 2024 Apr;114:106234. doi: 10.1016/j.clinbiomech.2024.106234. Epub 2024 Apr 3. PMID 38582028
- [Derived] Pechstein AE, Gollie JM, Keyser RE, Guccione AA. Walking Endurance and Oxygen Uptake On-Kinetics in Individuals With Parkinson Disease Following Overground Locomotor Training. J Neurol Phys Ther. 2023 Apr 1;47(2):99-111. doi: 10.1097/NPT.0000000000000423. Epub 2022 Dec 19. PMID 36538418
- See also: Supporting literature for performance and perceived fatigability — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3419324/